CLINICAL TRIAL: NCT02924545
Title: Evaluation of Osteoporosis Support After a Severe Osteoporotic Fracture in Women Over 50 Years in University Hospital
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2015/CGV-01
Record Dates: First submitted 2016-09-13; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-09

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluate the support of osteoporosis in women over 50 years with severe osteoporotic fractures (hip, vertebral, rib, Humeral, pelvic fractures) in the Nîmes University Hospital taking prediction of treatment of osteoporosis as criterion.

ELIGIBILITY:
Inclusion Criteria:

* patients over 50 years (> 50 years) with severe osteoporotic fractures (hip, vertebral, rib, Humeral, pelvic fractures) hospitalized in the Nîmes University Hospital

Exclusion Criteria:

* patient under 50 years
* Non osteoporotic fractures

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients over 50 years (> 50 years) hospitalized at the CHU de Nîmes all services (rheumatology , orthopedic surgery, emergency medicine versatile , physical medicine and rehabilitation, etc.) taken into charge between 1 January 2014 and 31 December 2014 for a wrist fracture , femoral neck or spine osteoporotic fracture.
  Patients supported for a fracture may be osteoporotic, will be identified using the PMSI (Programme de Médicalisation des Systèmes d'Information) data.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Is the treatment of osteoporosis scheduled according to the hospital report? yes/no | 1 year

IPD SHARING:
Plan to Share IPD: No